CLINICAL TRIAL: NCT01949233
Title: A Randomised, Double-blind, Placebo-controlled Pilot Trial of Irbesartan, Doxycycline and a Combination on Markers of Vascular Dysfunction in the Marfan Syndrome, Using Cardiovascular Magnetic Resonance Imaging
Brief Title: The Oxford Marfan Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-023612-14
Record Dates: First submitted 2013-08-06; First posted 2013-09-24 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Marfan Syndrome
MeSH Terms: conditions — Marfan Syndrome | interventions — Irbesartan; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Irbesartan 150-300mg (and doxycycline placebo) (Experimental): Irbesartan 150-300mg capsules daily for 6 months Doxycycline placebo capsules daily for 6 months
  Interventions: Drug: Irbesartan 150-300mg capsules daily for 6 months; Drug: Doxycycline placebo capsules daily for 6 months
- Doxycycline 100-200mg (and irbesartan placebo) (Experimental): Doxycycline 100-200mg capsules daily for 6 months Irbesartan placebo capsules daily for 6 months
  Interventions: Drug: Doxycycline 100-200mg capsules daily for 6 months; Drug: Irbesartan placebo capsules daily for 6 months
- Irbesartan 150-300mg and doxycycline 100-200mg (Experimental): Irbesartan 150-300mg capsules daily for 6 months Doxycycline 100-200mg capsules daily for 6 months
  Interventions: Drug: Irbesartan 150-300mg capsules daily for 6 months; Drug: Doxycycline 100-200mg capsules daily for 6 months
- irbesartan and doxycycline placebo (Placebo Comparator): Irbesartan placebo capsules daily for 6 months Doxycycline placebo capsules daily for 6 months
  Interventions: Drug: Doxycycline placebo capsules daily for 6 months; Drug: Irbesartan placebo capsules daily for 6 months

INTERVENTIONS:
Drug: Irbesartan 150-300mg capsules daily for 6 months
  Arms: Irbesartan 150-300mg (and doxycycline placebo); Irbesartan 150-300mg and doxycycline 100-200mg
Drug: Doxycycline 100-200mg capsules daily for 6 months
  Arms: Doxycycline 100-200mg (and irbesartan placebo); Irbesartan 150-300mg and doxycycline 100-200mg
Drug: Doxycycline placebo capsules daily for 6 months
  Arms: Irbesartan 150-300mg (and doxycycline placebo); irbesartan and doxycycline placebo
Drug: Irbesartan placebo capsules daily for 6 months
  Arms: Doxycycline 100-200mg (and irbesartan placebo); irbesartan and doxycycline placebo

SUMMARY:
The primary objective of the trial is to estimate the effects of allocation to irbesartan, or doxycycline, or a combination of both irbesartan and doxycycline, compared with placebo, on measures of elastic function of the aorta in people with the Marfan syndrome and enlargement of the aorta.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 13 years or above at last birthday (note that there is no upper age limit for inclusion in this trial)
* For those aged greater than or equal to 16 years of age at the time of enrolment, participant is willing and, in the opinion of the investigator, able to give informed consent for participation in the trial
* For those aged 13-15 at the time of enrolment, participant is willing and, in the opinion of the investigator, able to give informed assent, and parent/guardian is willing and able to give informed consent for participation in the trial.
* Weight ≥ 50kg
* Diagnosed with Marfan syndrome according to the revised Ghent criteria 1996
* Dilated aorta (BSA-adjusted aortic root z-score ≥2 at the aortic sinuses of Valsalva, using the method of Roman et al, or an absolute aortic root dimension >4.0cm at the sinuses of Valsalva measured using either echocardiography or CMR)
* If the participant is a female of child-bearing potential, they are willing to ensure effective contraception as defined in the contraception policy
* If the participant is taking β-blocker therapy, they are willing to stop taking these one week prior to each CMR scan
* Willing and, in the investigator's opinion, able to comply with all trial requirements
* Willing to allow his or her General Practitioner and if appropriate, Consultant, to be informed of his or her participation in the trial and of any clinical findings or issues which may arise

Exclusion Criteria:

* Female who is pregnant
* Female who is planning pregnancy within 6 months of enrolment
* Female who is breast feeding
* Previous aortic dissection
* Previous aortic surgery
* Bicuspid or unicuspid aortic valve
* Scheduled elective cardiac or aortic surgery within 6 months of enrolment
* Definite diagnosis of Loeys-Dietz or Shpritzen-Goldberg syndrome
* Known bilateral renal artery stenosis or renal artery stenosis to a single functioning kidney
* History of idiopathic intracranial hypertension
* Exposure to angiotensin receptor antagonists, angiotensin converting enzyme inhibitors, or medications containing these compounds in the 3 months prior to enrolment in the trial
* Absolute indication for angiotensin receptor antagonists, angiotensin converting enzyme inhibitors, doxycycline or other antibiotics of the tetracycline class at enrolment
* Taking β-blocker therapy for an indication other than the Marfan syndrome
* Participant has participated in another research study involving an investigational medicinal product or device in the 3 months prior to enrolment
* Renal impairment of a moderate or severe degree (eGFR <60 mls/min/1.73m2)
* Hyperkalaemia (>5.1 mmol/L)
* Significant hepatic impairment (ALT or AST >3 times upper limit of normal)
* History of allergic reaction or any other clinically significant intolerance to irbesartan or its constituents; other angiotensin receptor blockers / antagonists; angiotensin converting enzyme inhibitors, doxycycline or its constituents, or placebo medications or its constituents
* Contra-indications to MRI (e.g. implantable cardiac electronic device, claustrophobia, intracranial aneurysm clips and metallic ocular foreign bodies etc.)
* Participant currently required to take or likely to be required to start, in the 6 months following enrolment, a medicinal product which is known or suspected to interact, to a clinically significant extent, with irbesartan including: potassium supplementation, potassium sparing diuretics, lithium, regular use of antacids containing aluminium magnesium hydroxide
* Participant currently required to take or likely to be required to start, in the 6 months following enrolment, a medicinal product which is known or suspected to interact, to a clinically significant extent, with doxycycline including ergotamine and methysergide. This includes drugs known to induce the cytochrome P450 system to a clinically significant extent, including but not limited to, carbamazepine, phenytoin, rifampicin, griseofulvin, barbiturates or sulphonylureas.
* Alcohol dependence
* Any other significant disease, disorder or circumstance (e.g. terminal illness), which, in the opinion of the Investigator, may either put the participant at risk in the trial, or may introduce significant bias to the trial, or may affect the participant's ability to participate in the trial

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change (i.e. difference between first and last study visits) in aortic distensibility in the ascending aorta between allocation arms measured using CMR | 0 months and 6 months

SECONDARY OUTCOMES:
1. Change in aortic distensibility in the proximal and distal descending aorta between allocation arms measured using CMR | 0 and 6 months
2. Change in aortic dimensions in the proximal and distal descending aorta | 0 and 6 months
3. Change in mean and peak axial and mean and peak circumferential aortic wall shear stress between allocation arms estimated by CMR using a 4D flow sequence | 0 and 6 months
4. Change in peripheral (brachial) blood pressure between allocation arms measured using a calibrated, validated automated sphygmomanometer | 0 and 6 months
5. Change in central blood pressure, and augmentation index between allocation arms measured by applanation tonometry and by oscillometric sphygmomanometry | 0 and 6 months
6. Change in left ventricular volumes, mass and systolic function between allocation arms to placebo measured by CMR | 0 and 6 months
7. Change in aortic pulse wave velocity between allocation arms measured by CMR | 0 and 6 months
8. Change in carotid-femoral pulse wave velocity between allocation arms compared to placebo measured by applanation tonometry | 0 and 6 months
9. Change in TGF-β level, or other biomarker, between allocation arms compared to placebo | 0 and 6 months
10. Tolerability and safety of irbesartan and doxycycline, assessed by incidence of adverse reactions and change in health status score, using the SF-36 questionnaire | 0, 0.5 and 6 months
11. Document the frequency of aortic dissection, death from cardiovascular causes, or need for aortic root or valve surgery (if any) in each allocation arm | 0-6 months

CONTACTS AND LOCATIONS:
Overall Officials: J Colin Forfar, BSc (hons), MA(Oxon), MD, PhD,, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - University of Oxford, Oxford, Oxfordshire